CLINICAL TRIAL: NCT00048399
Title: Phase I/II Study of Allogeneic Stem Cell Transplantation For Patients With Graft Failure Following Allogeneic Transplantation Using MHC Identical or Near Identical Donors and Submyeloablative Conditioning With CAMPATH 1H (CAMGRAFT)
Brief Title: Stem Cell Transplantation for Patients With Graft Failure Following an Allogeneic Transplant, Using Identical or Near Identical Donors and Less Toxic Conditioning With CAMPATH 1H
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: accrual was slow
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Robert Krance, Professor, Baylor College of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H9446; CAMGRAFT
Record Dates: First submitted 2002-10-30; First posted 2002-11-01 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Graft Failure
MeSH Terms: interventions — fludarabine; Alemtuzumab; Tacrolimus; Stem Cell Transplantation

INTERVENTIONS:
Drug: Fludarabine
Drug: CAMPATH 1H
Drug: FK506
Procedure: Stem Cell Transplantation

SUMMARY:
To assess the safety, feasibility, and rate of donor engraftment for patients with primary or secondary engraftment failure after treatment with fludarabine and CAMPATH 1H used as a preparative regimen for HLA-identical sibling blood stem cell transplantation (SCT).

To assess the safety, feasibility, and rate of donor engraftment for patients with primary or secondary engraftment failure after treatment with fludarabine and CAMPATH 1H as a preparative regimen for matched unrelated or single antigen mismatched family donor marrow transplantation.

DETAILED DESCRIPTION:
Study participants will receive the following treatment:

Day -5 to -2...Fludarabine 30mg/m2* and CAMPATH** 1H 10mg IV

Day -1.........Day of rest

Day 0..........Stem cell transplant (infusion)

Where possible, patients will receive peripheral blood stem cells. When peripheral stem cells are unavailable (e.g. from some unrelated donor centers) or insufficient, bone marrow will be substituted. If peripheral blood stem cell collection is performed, the donor will be stimulated with G-CSF for 5 days and cells collected and frozen until the stem cell target number is obtained prior to the patient beginning the therapy. If a bone marrow harvest is performed, this will be performed on Day 0 (infusion day). After transplantation, G-CSF 5 micrograms/kg/day will be administered SC from day 7 until granulocytes >1000/ul.

Because CAMPATH-1H infusions will provide a persisting level of antibody over the transplant period, it will contribute to anti-GvHD activity. Additional GVHD prophylaxis will consist of FK506 administered IV via continuous infusion over 24 hours from Day-2 until engraftment or when the patient is able to take by mouth, every 12 hours. This is continued until 6 months post-transplantation. The dose is then tapered every 2 weeks until discontinued. All patients will receive supportive care (prophylaxis for antimicrobial, antiviral, antifungal and Pneumocystis Pneumonia, transfusions of blood products and intravenous gamma globulin and routine laboratory testing of chemistry and complete blood counts) as per Cell and Gene Therapy Standard Operating Procedures (SOP).

Donor engraftment will be evaluated via standard bone marrow studies (cytogenetics/DNA studies for chimerism) on days 30, 60, 100, 180 and 365 post transplantation. If these studies reveal loss of donor cells on two consecutive studies and/or evidence of relapsing disease, the donor will undergo a peripheral blood stem cell harvest via G-CSF stimulation.

ELIGIBILITY:
INCLUSION CRITERIA

* Diagnosis of engraftment failure either primary or secondary, following allogeneic transplantation. Graft failure is defined as absolute neutrophil count < 500/mm3 and/or platelet count < 20,000/mm3. Primary graft failure is defined as failure to maintain absolute neutrophil count > / = 500/mm3 for 3 consecutive days following allogeneic transplantation. Secondary graft failure is defined as failure to sustain an absolute neutrophil count > / = 500/mm3 after attainment of primary engraftment or failure to sustain platelet count > / = 20,000/mm3 despite neutrophil engraftment. For SCID patients, graft failure is defined as failure to recover > / = 500/mm3 T-cells and/or failure to generate satisfactory response to in vitro mitogen stimulation. For patients with genetic diseases, engraftment failure is defined as donor chimerism insufficient to correct or overcome the genetic or metabolic deficiency.
* Available Healthy Donor without any contraindications for donation (5/6 or 6/6 related donor or 5/6 or 6/6 unrelated donor (molecular typing for DRB1)
* Age between birth and 65
* For women of childbearing potential, negative pregnancy test

EXCLUSION CRITERIA

* Pregnant and lactating women or women unwilling to use contraception.
* Uncontrolled intercurrent infection
* Refractory AML or ALL
* Untreated Blast Crisis for CML
* Uncontrolled High-grade lymphoproliferative disease/lymphoma
* Unstable angina and uncompensated congestive heart failure (Zubrod of 3 or greater)
* Severe chronic pulmonary disease requiring oxygen (Zubrod of 3 or greater)
* Hemodialysis dependent
* Active Hepatitis or cirrhosis with total bilirubin, SGOT, or SGPT greater than 3 x normal.
* Concurrent solid organ malignancy not in remission, except for Stage 0 or A prostate cancer.
* Unstable Cerebral vascular disease and recent hemorrhagic stroke (less than 6 months)
* Active CNS disease from hematological disorder.

Max Age: 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40
Dates: Start 2000-12; Primary Completion 2003-10-31 (Actual); Study Completion 2003-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert K. Krance, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Texas Children's Hospital, Houston, Texas
  - The Methodist Hospital, Houston, Texas